CLINICAL TRIAL: NCT06135909
Title: CHina Registry for the chAracteristics and Management strategieS of patiEnts With Pulmonary Hypertension Using Targeted Therapy
Brief Title: CHASE Registry of Patients With Pulmonary Hypertension Receiving Targeted Therapy
Status: Recruiting | Type: Observational
Sponsor: Chinese Pulmonary Vascular Disease Research Group (Other)
Responsible Party: Sponsor
Other Study IDs: CHASE
Record Dates: First submitted 2023-11-12; First posted 2023-11-18 (Actual); Last update posted 2024-01-18 (Actual); Status verified 2023-11

CONDITIONS: Pulmonary Hypertension
MeSH Terms: conditions — Hypertension, Pulmonary

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- PH Patients receiving targeted drugs treatment: Patients with pulmonary hypertension receiving targeted drugs treatment

SUMMARY:
CHina Registry for the chAracteristics and Management strategieS of patiEnts With Pulmonary Hypertension Using Targeted Therapy (CHASE Study)

DETAILED DESCRIPTION:
The purpose of this study was to establish the clinical characteristics and treatment strategies of targeted pulmonary hypertension patients in China: a multicenter, prospective case registry (CHASE) study to describe the clinical characteristics, treatment used, disease progression, and outcomes (e.g., death, hospitalization) of patients taking targeted drugs in real-world clinical practice. This study will collect high-quality real-world data that can be used as a standalone dataset or combined with other data sources to address critical issues in the PH field.

This is a prospective, observational, multicenter study. The expected number of enrolled cases for the entire study: at least 5000; No experimental group and control group were divided. Patients were followed up every 6 months ±2 weeks after enrollment for 3 years. The study selected patients who signed informed consent, aged 18-25 years, clinically diagnosed with pulmonary hypertension, and were applying or planning to apply targeted drugs for pulmonary hypertension as the study objects. The primary endpoint was the incidence of clinical exacerbations at 1 year after enrollment. Secondary endpoints were all-cause mortality at 1, 2, and 3 years after enrollment, rate of lung transplantation or combined cardiopulmonary transplantation, 6-minute walking distance, NT-proBNP level, WHO cardiac function grade, ratio of right ventricular end-diastolic diameter to left ventricular end-diastolic diameter, pulmonary hypertension targeted drug regimen, and incidence of associated adverse reactions.

ELIGIBILITY:
Inclusion Criteria:

* Sign informed consent;
* Between the ages of 18 and 85;
* Clinical diagnosis of pulmonary hypertension, using or planning to use pulmonary hypertension targeted drugs (including any one or more of the following: prostacyclin analogues, endothelin receptor antagonists, phosphodiesterase inhibitors, soluble guanylate cyclase agonists and prostacyclin receptor agonists).

Exclusion Criteria:

* Have a history of mental illness or drug or poison addiction, and can not sign informed consent or can not cooperate with the experimental study;
* Patients with malignant tumor and other diseases and life expectancy of less than half a year;
* Short-term (less than 2 weeks) patients taking targeted drugs for pulmonary hypertension

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with pulmonary hypertension receiving targeted therapy
Sampling Method: Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of clinical worsening events 1 year after enrollment | 1 year after enrollment
  All-cause death, Pulmonary hypertension progression associated with re-hospitalization, Progress of pulmonary hypertension disease

SECONDARY OUTCOMES:
Incidence of all-cause death 1,3,5 year(s) after enrollment | 1,3,5 year(s) after enrollment
  Incidence of all-cause death 1,3,5 year(s) after enrollment

CONTACTS AND LOCATIONS:
Overall Officials: Zhihong Liu, M.D., Ph.D, Principal Investigator — Chinese Academy of Medical Sciences, Fuwai Hospital
Locations (1):
- Center for Respiratory and Pulmonary Vascular Diseases, Fuwai hospital, CAMS & PUMC, Beijing, China